CLINICAL TRIAL: NCT06449963
Title: The Effect of Health Belief Model-Based Education on Daily Water Consumption and Dehydration Symptoms in Elderly Individuals Who Do Not Drink Enough Water
Brief Title: Effect of Health Belief Model Education on Water Intake in the Elderly (HBM-Water Study)
Acronym: HBM-Water Stud
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bayburt University (Other)
Collaborators: Ataturk University (Other)
Responsible Party: Principal Investigator, Arzu ÇİMEN, PhD Candidate (Doctoral Student), Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ATAUNI-NURS-FON-2024; ATAUNI-BAPSIS-TDK-2024-13931 (Other Grant/Funding Number: Atatürk University Scientific Research Projects (BAP) Support); BAYBU-IRB-2024-14 (Other: Bayburt University Non-invasive Clinical Research Ethics Committee Approval, dated 23.02.2024, Decision Number 2024/14)
Record Dates: First submitted 2024-06-04; First posted 2024-06-10 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Dehydration; Water Consumption in Elderly
Keywords: Health Belief Model; Elderly; Hydration; Education Program
MeSH Terms: conditions — Dehydration

STUDY DESIGN:
Intervention Model Description: This study uses a parallel assignment model where participants are randomly assigned to either the intervention group or the control group. The intervention group will receive the Health Belief Model (HBM)-based education program, while the control group will receive no education. The purpose is to compare the effectiveness of the HBM-based education program on increasing daily water consumption among elderly individuals.
Masking Description: There are no additional masked parties in this clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health Belief Model Education Group (Experimental): Participants in this arm will receive a structured educational program aimed at increasing their daily water intake. The program is based on the principles of the Health Belief Model (HBM) and includes the following components:
  Educational Sessions: Weekly group sessions led by trained health educators, focusing on the importance of hydration, the benefits of adequate water intake, and strategies to incorporate more water into daily routines.
  Behavioral Strategies: Practical tips and techniques to overcome barriers to water intake, such as setting daily water goals, using water bottles, and incorporating water-rich foods into the diet.
  Personalized Feedback: Individualized feedback and support provided through weekly one-on-one meetings with a health coach to track progress and address any challenges.
  Educational Materials: Distribution of printed and digital materials, including pamphlets and interactive tools, to reinforce learning and support behavior change.
  Interventions: Behavioral: Health Belief Model Education
- No Education Control Group (No Intervention): Participants in this arm will not receive any specific education or intervention and will follow their usual routines. This group will serve as a control to compare the effectiveness of the Health Belief Model-based education program administered to the intervention group. The daily water intake of participants in this group will be recorded using standardized intake diaries, and averages will be calculated weekly.

INTERVENTIONS:
Behavioral: Health Belief Model Education — Participants in this group will receive a structured training program with the aim of increasing daily water consumption and reducing symptoms of dehydration. The program is based on the principles of the Health Belief Model and includes the following components:
  Initial and mid-Program training: Will be conducted by a trained health educator, each lasting 60 minutes. Two weeks after the first training, the same training will be given again for reinforcement purposes.
  Session Content: Covers the importance of hydration, strategies to increase water intake (using reminders, setting goals, integrating water-rich foods), and the health benefits of adequate hydration (e.g., improved cognitive function, better physical health).
  Training Materials: Booklet prepared for training. Behavioral Strategies: Practical tips for overcoming barriers to drinking more water, such as setting daily water intake goals and using diaries to track progress.
  Arms: Health Belief Model Education Group

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a Health Belief Model (HBM)-based education program to increase daily water consumption among elderly individuals aged 65 and above. Participants will be divided into two groups; one group will receive HBM-based education, and the other group will not receive any education. The effects of the education program on daily water consumption and dehydration symptoms will be assessed.

DETAILED DESCRIPTION:
The study has a randomized controlled design and will last 1 month. The study group will be given a Health Belief Model (HBM)-based training program for 1 month, and the same training will be given again after 2 weeks to reinforce the training, while the control group will not receive any training. Participants; Daily water consumption will be collected and dehydration symptoms will be evaluated at baseline and at the end of 1 month, and differences between groups will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

Aged 65 years and older. Consuming less than 1000 ml of water daily.

Exclusion Criteria:

Scoring below 17 on the Mini-Mental State Examination. Being bedridden. Having a medical condition that requires fluid restriction. Taking diuretic medications.

Withdrawal Criteria:

Elderly participants who wish to withdraw from the study at any stage of the research process.

Participants who meet the exclusion criteria during the study period.

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Average Daily Water Intake (liters) | Data collection at baseline, 24-hour intervals, and daily data collection until the end of 30 days
  In order to determine the effect of providing health belief model education on the level of water consumption; The daily water consumption amount is determined before training. After the training, they are asked to record the amount of water they will consume daily for 30 days on the record chart. Then, the amount of water consumed at 3-day intervals is called and recorded by the patient. The amount of change in daily water consumption at the end of 30 days will determine the effect level of the training.

SECONDARY OUTCOMES:
Change in Hydration Status (urine specific gravity) | At baseline, after 15 days, and on day 30
  In order to determine the effect of providing health belief model education on the change in hydration status; Before training, the specific gravity of the urine is measured using a refractometer. The same measurement is repeated 15 days later, after reinforcement training, and on the 30th day of the study. In this way, the effect of training on the change in hydration status will be determined.

CONTACTS AND LOCATIONS:
Locations (1):
- Atatürk University Health Sciences Institute, Department of Nursing Principles, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
When I answered yes, the system accepted the URL I gave as incorrect, so I chose the no option to continue.
  Time Frame: "IPD and supporting information will be available for 3 years, starting 6 months after the article is published."
  Access Criteria: "Researchers who present a methodologically sound proposal will have access to the IPD and supporting information. To gain access to the data, those requesting data will be required to sign a data access agreement. Suggestions should be directed to [arzucimen@bayburt.edu.tr]." https://www.atauni.edu.tr/

REFERENCES:
- [Background] Ciftci B, Yildiz GN, Avsar G, Kose S, Aydin E, Dogan S, Celik S. Development of the Thirst Discomfort Scale: A Validity and Reliability Study. Am J Crit Care. 2023 May 1;32(3):176-183. doi: 10.4037/ajcc2023954. PMID 37121897
- See also: Development of the Thirst Discomfort Scale: A Validity and Reliability Study — https://pubmed.ncbi.nlm.nih.gov/37121897/